CLINICAL TRIAL: NCT05992168
Title: A Prospective, Multicenter, Single Arm Clinical Trial to Evaluate the Safety and Efficacy of Pulmonary Artery Thrombectomy Devices for the Treatment of Acute Pulmonary Embolism
Brief Title: Stent-Retriever for Acute Massive Pulmonary Embolism (SRAME)
Acronym: SRAME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical trial was terminated ahead of schedule due to strategic changes within the company.
Sponsor: Suzhou Zenith Vascular Scitech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZZT-CP-202301
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: PE - Pulmonary Embolism; PE - Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stent-Retriever arm (Experimental): Device: Stent-Retriever
  Interventions: Device: Stent-Retriever

INTERVENTIONS:
Device: Stent-Retriever — all the participants in this group will be performed with Stent-Retriever

SUMMARY:
To evaluate treatment outcomes of patients diagnosed with pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

- 1.18≤ age ≤75, no gender limitation; 2.patients clinically diagnosed as acute pulmonary embolism requiring pulmonary artery thrombosis clearance; 3.RV/LV ratio ≥0.9; 4.Patients who agreed to participate in the study and voluntarily signed the informed consent.

Exclusion Criteria:

1. Patients with systolic blood pressure<90 mmHg and lasting for 15 minutes or requiring maintenance of systolic blood pressure ≥ 90 mmHg;
2. Patients with known severe pulmonary hypertension;
3. Patients with Hematocrit <28%;
4. Patients with known structural heart disease;
5. Patients with left bundle branch block;
6. Patients with history of chronic left heart failure and left ventricular ejection fraction ≤30%;
7. Patients with abnormal renal function (serum creatinine > 1.8 mg/dL or >159 umol/L);
8. Patients with known coagulopathy or bleeding tendency (platelet <100×109/L, or INR> 3);
9. Patients who cannot receive antiplatelet or anticoagulant therapy;
10. Patients who underwent cardiovascular or pulmonary open surgery within 7 days before peocedure;
11. Patients with intracardiac thrombosis;
12. Patients treated with extracorporeal membrane oxygenation;
13. Patients known to be allergic to contrast agents;
14. Patients with diseases that may cause difficulty in treatment or evaluation (such as malignant tumor, acute infectious disease, sepsis, general condition that cannot tolerate procedure, life expectancy less than one year, etc.);
15. Females who are pregnant or in lactation;
16. Patient is currently enrolled in another investigational study protocol;
17. Other conditions not suitable for inclusion judged by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Reduction in RV/LV ratio from baseline to 48 hours | 48 hours post procedure
  Endpoint events will be assessed from the time of treatment of the pulmonary embolism through hospital discharge, or through 48 hours post treatment, whichever comes first.
Major Adverse Events from baseline to 48 hours | 48 hours post procedure
  Endpoint events will be assessed from the time of treatment of the pulmonary embolism through hospital discharge, or through 48 hours post treatment, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No